CLINICAL TRIAL: NCT01429116
Title: An Extension Open-Label Safety Study of a 24-month 20 mg Dose Regimen of Tasimelteon for the Treatment of Non-24-Hour Sleep-Wake Disorder (N24HSWD) in Blind Individuals With no Light Perception Who Have Enrolled in Other Tasimelteon Clinical Trials
Brief Title: Tasimelteon for the Treatment of Non-24-hour Sleep-Wake Disorder (N24HSWD) in Blind Individuals With no Light Perception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VEC-162-3204
Record Dates: First submitted 2011-08-30; First posted 2011-09-05 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Non-24-Hour Sleep-Wake Disorder
Keywords: Blindness; Eye Diseases; Nap Disorders; Circadian Rhythm Disorders; Sleep Disorders; Circadian Rhythm Sleep Disorders; Dyssomnias; Nervous System Diseases
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Blindness; Eye Diseases; Chronobiology Disorders; Sleep Wake Disorders; Dyssomnias; Nervous System Diseases | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tasimelteon (Experimental): 20 mg tasimelteon capsules, PO daily for 24 months + 12 month optional extension
  Interventions: Drug: tasimelteon

INTERVENTIONS:
Drug: tasimelteon — 20 mg tasimelteon capsules, PO daily for 24 months + 12 month optional extension
  Other Names: VEC-162

SUMMARY:
The purpose of this study is to evaluate the safety of tasimelteon in male and female patients who suffer from Non-24-Hour Sleep-Wake Disorder.

DETAILED DESCRIPTION:
Non-24-Hour Sleep-Wake Disorder (N24HSWD) occurs when individuals are unable to synchronize their endogenous circadian pacemaker to the 24-hour light-dark cycle, and the timing of their circadian rhythm instead reflects the intrinsic period of their endogenous circadian pacemaker. As a result, the circadian rhythm of sleep-wake propensity in these individuals moves gradually later and later each day if there circadian period is > 24 hours and earlier and earlier is < 24 hours. These individuals will be able to sleep well at night when their sleep-wake propensity rhythm is approximately aligned with the 24-hour light-dark and social cycle. However, after a short time, the endogenous sleep-wake propensity rhythm and the 24-hour light-dark cycle will move out of synchrony with each other, and they may have difficulty falling asleep until well into the night. In addition to problems sleeping at the desired time, the subjects experience daytime sleepiness and daytime napping. As time progresses, the endogenous circadian rhythm of sleep-wake propensity in these individuals moves further and further away from the 24-hour light-dark cycle and gradually, these individuals are unable to sleep at night and as a result experience extreme sleepiness during the daytime hours and more frequent naps with a longer duration. Eventually, the sleep-wake time moves back into alignment with the social time for sleep and the individuals sleep well at night and have decreased daytime napping. The alignment between their endogenous circadian rhythms and the 24-hour day is temporary as they are continually drifting later and later each day.

The study is comprised of one 24-month treatment phase, as all subjects enrolled in the trial have already been diagnosed with N24HSWD. Frequency of study visits will depend on the subject's prior length of exposure to tasimelteon; accordingly, subjects will be assigned to one of two groups upon enrollment into the study. The short-term exposure group will consist of subjects for which it is possible at screening that they have been exposed to tasimelteon for less than 6 months. The long-term exposure group will consist of subjects who have more than 6 months of exposure to tasimelteon.

After completion of the 24-month treatment phase, subjects have the option to enroll into the optional open-label extension sub-study for an additional 52 weeks. Frequency of visits will be identical regardless of previous exposure (short term/long term).

ELIGIBILITY:
Inclusion Criteria:

1. Ability and acceptance to provide informed consent;
2. Men or women at least 18 years of age or older who meet one of the following:

   * Has enrolled in VP-VEC-162-3201 (with sponsor approval)
   * Has completed VP-VEC-162-3203
   * Was deemed a non-responder in VP-VEC-162-3203
   * Has enrolled in VP-VEC-162-3203 (with sponsor approval)
   * Has a previous diagnosis of N24HSWD
   * The subject is totally blind and meets the following Diagnostic and Statistical Manual of Mental Disorders 5 diagnostic criteria

     * A persistent or recurrent pattern of sleep disruption that is primarily due to an alteration of the circadian system or to a misalignment between the endogenous circadian rhythm and the sleep-wake schedule required by an individual's physical environment or social or professional schedule.
     * The sleep disruption leads to excessive sleepiness or insomnia, or both.
     * The sleep disturbance causes clinically significant distress or impairment in social, occupational, and other important areas of functioning.

   Specifically: A pattern of sleep-wake cycles that is not synchronized to the 24-hour environment, with a consistent daily drift (usually to later and later times) of sleep onset and wake times.
3. For US participants only: Males, non-fecund females (i.e., surgically sterilized,if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing during the study and for one month following the last dose and must have a negative pregnancy test at the screening and baseline visits Note: Women using hormonal methods of birth control must use an additional method of birth control during the study and for one month after the last dose.
4. Diagnosis of N24HSWD in a previous tasimelteon study;
5. Willing and able to comply with study requirements and restrictions;

Exclusion Criteria:

1. History (within the 12 months prior to screening) of psychiatric disorders including Major Depressive Disorder, Generalized Anxiety Disorder, Axis II Disorders, delirium or any other psychiatric disorder that in the opinion of the clinical investigator would affect participation in the study or full compliance with study procedures;
2. History of intolerance and/or hypersensitivity to melatonin or melatonin agonists;
3. History of drug or alcohol abuse as defined in DSM-IV, Diagnostic Criteria for Drug and Alcohol Abuse, within the 12 months prior to screening and/or regular consumption of alcoholic drinks (> 40g/day);
4. Patients having any current suicidal ideation of type 4 or 5 on the C-SSRS at Screening or Baseline;
5. Patient is at risk of suicide, in the opinion of the Investigator. Evidence of suicide risk could include any suicide attempt within the past year or any other suicidal behavior within the past year;
6. Current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction unless currently controlled and stable;
7. Clinically significant deviation from normal in vital signs measurements, or physical examination findings at screening or baseline as determined by the clinical investigator;
8. Pregnant or lactating females;
9. Smoke more than 10 cigarettes/day;
10. Exposure to any investigational drug other than tasimelteon, including placebo, within 30 days, 5 half-lives, or the exclusion period given by a previous study in which the patient has participated in, whichever of the three scenarios is longer.
11. Unwilling or unable to discontinue usage of medication listed in Section 8.2.1;
12. Any other sound medical reason as determined by the clinical investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (AEs) | 24 months + 12 month optional extension
  Treatment-emergent adverse events will be summarized by presenting the number and percentage of patients having any treatment-emergent AE, having an AE in each body system, and having each individual AE.

SECONDARY OUTCOMES:
Number of participants with changes in Clinical Laboratory Data | 24 months + 12 month optional extension
  Standard Serum Hematology and Chemistry tests will be performed at baseline and through the 24 months of treatment
Number of participants with newly occurring or worsening ECG abnormalities | 24 months + 12 month optional extension
Number of participants with clinically notable Vital Signs and Body Measurements | 24 months + 12 month optional extension
Number of participants who report a positive result for the Columbia Suicide Severity Rating Scale (C-SSRS) | 24 months + 12 month optional extension

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (22):
- United States (22):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - SDS Clinical Trials Inc., Orange, California
  - VA Palo Alto Health Care System/PAIRE (San Fransisco Bay Area), Palo Alto, California
  - St. Johns Sleep Disorder Center - St. Johns Medical Plaza, Santa Monica, California
  - Radiant Research - Denver, Denver, Colorado
  - PAB Clinical Research Inc., Brandon, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Sleep Disorders Center Of Georgia, Atlanta, Georgia
  - Suburban Lung Associates SC (Chicago Metropolitan Area), Elk Grove Village, Illinois
  - The Center for Sleep and Wake Disorders (Washington, D.C. Metropolitan Area), Chevy Chase, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Head-Pain Neurological Institute, Ann Arbor, Michigan
  - St. Luke's Sleep Medicine and Research Center (St. Louis Metropolitan Area), Chesterfield, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Ohio Sleep Medicine Institute (Columbus Metropolitan Area), Dublin, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Columbia Research Group Inc., Portland, Oregon
  - Center for Sleep Medicine at Chestnut Hill Hospital, Philadelphia, Pennsylvania
  - Consolidated Clinical trials, Pittsburgh, Pennsylvania
  - SleepMed, Inc. - Columbia, Columbia, South Carolina
  - Todd J. Swick, M.D., P.A., Houston, Texas